CLINICAL TRIAL: NCT04549506
Title: The Hypothesis of Emotional Empathy Imbalance in Autism: Conscious and Non-conscious Processing of Emotional Faces
Brief Title: Autism, Emotional Processing, and the Amygdala
Status: Completed | Type: Observational
Sponsor: Yawei Cheng (Other)
Responsible Party: Sponsor-Investigator, Yawei Cheng, Professor, National Yang Ming Chiao Tung University
Organization: National Yang Ming Chiao Tung University (Other)
Other Study IDs: YM102035
Record Dates: First submitted 2017-09-20; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ASD group: There is no intervention to be administered in this study. Here, this fMRI study used the backwardly masked paradigm to elucidate how perceiving emotional expressions affects amygdala engagement and its related functional connectivity across two participant groups: ASD with and controls. All ASD participants were diagnosed using the Diagnostic and Statistical Manual of Mental Disorders 5th Edition's (DSM-5) diagnostic criteria (APA, 2013) and conﬁrmed by clinical consensus. ASD individuals were recruited from a community autism program and referred to children's health doctors and child psychiatrists. Exclusion criteria for all participants were neurological abnormalities, a history of epilepsy or seizures, head trauma and IQ <75. The subjects did not participate in any intervention or drug programs during the experimental period.
- Control group: There is no intervention to be administered in this study. Here, this fMRI study used the backwardly masked paradigm to elucidate how perceiving emotional expressions affects amygdala engagement and its related functional connectivity across two participant groups: ASD with and controls. The participants in the age- and sex-matched control group were recruited from the local community, and screened for major psychiatric illnesses by conducting structured interviews.

SUMMARY:
Empathy imbalance hypothesis suggests that individuals with autism Spectrum Disorder (ASD) should have a deficit of cognitive empathy and a surfeit of emotional empathy. Considering that inconsistent amygdala reactivity to emotional faces might be ascribed to aberrant attention in ASD, the investigators hypothesized to investigate if there would be an imbalance between conscious and nonconscious emotional processing. This fMRI study recruited 26 youths and young adults with autism spectrum disorder and 25 matched controls, and measured their amygdala reactivity and functional connectivity in response to conscious and nonconscious (backward masked) perception of threatening faces.

Keywords: Autism Spectrum Disorder; amygdala reactivity; emotional processing; fMRI

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of severity of Autism-Spectrum Disorders
* IQ > 75

Exclusion Criteria:

* Neurological abnormalities,
* A history of epilepsy or seizures, head trauma a
* IQ <75

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Autism group: 26 individuals with ASD meeting DSM-V criteria Control group: 25 gender, and age matched healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2014-04-19 (Actual); Primary Completion 2016-09-21 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Age | 1 minutes
  Age in years
Anxiety scores | 10 minutes
  State-Trait Anxiety Inventory (STAI)
Severity of Austism-Spectrum Disorders | 20 minutes
  Autism-Spectrum Quotient (AQ)
Color identification task | 10 minutes
  During fMRI scanning, subjects watched emotional faces and performed the color identification task, in which they were asked to judge the color of each face (pseudo-colored in either red, yellow, or blue) and to indicate the answer by a keypad button press.
Detection task | 10 minutes
  Immediately after fMRI scanning, participants underwent the detection task, during which they were shown all of the stimuli again and alerted of the presence of fearful faces. The subjects were administered a forced-choice test under the same presentation conditions as those during scanning and asked to indicate whether they observed a fearful face or not.
fMRI response | 10 minutes
  During fMRI scanning, subjects watched emotional faces and performed the color identification task, in which they were asked to judge the color of each face (pseudo-colored in either red, yellow, or blue) and to indicate the answer by a keypad button press.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liddell BJ, Williams LM, Rathjen J, Shevrin H, Gordon E. A temporal dissociation of subliminal versus supraliminal fear perception: an event-related potential study. J Cogn Neurosci. 2004 Apr;16(3):479-86. doi: 10.1162/089892904322926809. PMID 15072682
- [Background] Williams LM, Kemp AH, Felmingham K, Liddell BJ, Palmer DM, Bryant RA. Neural biases to covert and overt signals of fear: dissociation by trait anxiety and depression. J Cogn Neurosci. 2007 Oct;19(10):1595-608. doi: 10.1162/jocn.2007.19.10.1595. PMID 17854280
- [Background] Schumann CM, Amaral DG. Stereological analysis of amygdala neuron number in autism. J Neurosci. 2006 Jul 19;26(29):7674-9. doi: 10.1523/JNEUROSCI.1285-06.2006. PMID 16855095
- [Background] Eimer M, Kiss M, Holmes A. Links between rapid ERP responses to fearful faces and conscious awareness. J Neuropsychol. 2008 Mar;2(Pt 1):165-81. doi: 10.1348/174866407X245411. PMID 19330049
- [Background] Hall GB, Doyle KA, Goldberg J, West D, Szatmari P. Amygdala engagement in response to subthreshold presentations of anxious face stimuli in adults with autism spectrum disorders: preliminary insights. PLoS One. 2010 May 25;5(5):e10804. doi: 10.1371/journal.pone.0010804. PMID 20520836